CLINICAL TRIAL: NCT03346330
Title: An Exploratory, Randomised, Double-blind, Placebo-controlled, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food-effect of TRK-750 in Healthy Adults and Patients With Peripheral Neuropathic Pain
Brief Title: Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), Food-effect of TRK-750
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 750P1C01
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Healthy, Peripheral Neuropathic Pain
Keywords: Chronic pain; Neuropathic pain
MeSH Terms: conditions — Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRK-750, single and multiple doses (Experimental)
  Interventions: Drug: TRK-750
- Placebo, single and multiple doses (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRK-750 — TRK-750 capsule
  Arms: TRK-750, single and multiple doses
Drug: Placebo — Placebo capsule
  Arms: Placebo, single and multiple doses

SUMMARY:
This is an exploratory, randomised, double-blind, placebo-controlled, Phase I study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and food-effect of single and multiple, ascending oral doses of TRK-750 in healthy adults and patients with peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers
* Female subjects who are either:

  1. Non-childbearing potential, or permanently sterile OR
  2. Childbearing potential and agree to use at least one form of highly effective contraception
* Male subjects, with a female sexual partner of childbearing potential or a pregnant or breastfeeding partner, must agree to use barrier contraception (male condom) for the treatment period and for at least three months after the end of the systemic exposure of the study drug.
* Satisfactory medical assessment with no clinically significant or relevant abnormalities.
* Ability to provide written, personally signed, and dated informed consent.

Exclusion Criteria:

* Current or recurrent disease
* Current or relevant history of physical or psychiatric illness
* Positive test for Hepatitis B, Hepatitis C or human immunodeficiency virus antibody (HIV) at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events as assessed by CTCAE v4.03 | Up to 10-14days after last dose
Proportion of subjects with clinically significant changes in laboratory safety tests | Up to 10-14days after last dose
Proportion of subjects with morphological and/or rhythm abnormalities on electrocardiogram | Up to 10-14days after last dose
Proportion of subjects with clinically significant changes in electrocardiogram time intervals | Up to 10-14days after last dose
Proportion of subjects with clinically significant changes in vital signs:systolic blood pressure(mmHg) | Up to 10-14days after last dose
Proportion of subjects with clinically significant changes in vital signs:diastolic blood pressure(mmHg) | Up to 10-14days after last dose
Proportion of subjects with clinically significant changes in vital signs:pulse rate(bpm) | Up to 10-14days after last dose
Proportion of subjects with clinically significant changes in vital signs:body temperature(°C) | Up to 10-14days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- London, London, United Kingdom